CLINICAL TRIAL: NCT01165294
Title: Investigate the Effect of S-Ketamine, as Pharmacological Model of Schizophrenia, on the Attentiveness and Working Memory Simultaneously Measured With Functional Magnetic Resonance Imaging(fMRI)/Electroencephalogram(EEG)
Brief Title: The Effect of Ketamine on Attentiveness
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Director, Janssen Pharmaceutica N.V., Belgium
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: CR017368
Record Dates: First submitted 2010-07-15; First posted 2010-07-19 (Estimated); Last update posted 2010-08-06 (Estimated); Status verified 2010-08

CONDITIONS: Schizophrenia
Keywords: Ketamine
MeSH Terms: conditions — Schizophrenia | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 001 (Experimental): ketamine An intravenous bolus of 0.1 mg/kg will be given in 5 minutes followed by a 1 minute break after which a continuous infusion will start at 0.015625 mg/kg/min.
  Interventions: Drug: ketamine
- 002 (Experimental): Placebo An intravenous bolus will be given in 5 minutes time followed by a 1 minute break after which a continuous infusion will start. Dosage lowered every 10 minutes
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — An intravenous bolus will be given in 5 minutes time followed by a 1 minute break after which a continuous infusion will start. Dosage lowered every 10 minutes
  Arms: 002
Drug: ketamine — An intravenous bolus of 0.1 mg/kg will be given in 5 minutes followed by a 1 minute break after which a continuous infusion will start at 0.015625 mg/kg/min.
  Arms: 001

SUMMARY:
The objective of this study is to develop an exploratory design for future Proof-of-Concept trials which reliably and accurately measure the central nervous system (CNS) effects of potentially new drugs that oppose the effects of ketamine at a subanesthetic dose level given to healthy volunteers. A functional magnetic resonance imaging (fMRI) and electroencephalogram (EEG) performed simultaneously during a ketamine challenge will register the effects triggered by Ketamine.

DETAILED DESCRIPTION:
This will be a double-blind (neither physician nor patient knows the name of the assigned drug), placebo-controlled, randomized (study drug assigned by chance), 2 way crossover ketamine challenge study (participants may receive different interventions sequentially during the trial) in 24 healthy male volunteers. For all participants, this study will consist of an eligibility screening examination, two 2-day treatment periods, separated by at least 1 week, and a follow-up examination about 7 days after last dose administration. The maximal study participation for each volunteer will be around 6 weeks. Apart from observing possible neural and vascular ketamine effects, the cerebral ketamine effects will be investigated by simultaneously performing fMRI/EEG during ketamine administration. These investigations will be done while volunteers rest as well as during cognitive testing (visual oddball task). Safety evaluations include continuous monitoring of vital signs and oxygen saturation. Due to the pharmacokinetic properties of ketamine the assessments will start after an intravenous ketamine bolus (drug given directly into the vein over a short period of time) followed by a 1 minute break. During the assessments there is a continuous intravenous (minimal) drug administration. Before the assessments start there will be an intravenous bolus of 0.1 mg/kg ketamine in 5 minutes time followed by a 1 minute break after which a continuous infusion will start of 0.015625 mg/kg/min ketamine. Since the plasma level elevates during the infusion the administered dose will be lowered by 10% every 10 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Normal ECG and safety assessments, or minor no-relevant deviations, at screening
* Vital signs: systolic between 100 and 140 mmHg and diastolic between 50 and 90 mmHg and heart rate between 45 and 90 beats/min
* No medication intake in the last four weeks
* Volunteers must have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study and to adhere to the prohibitions and restrictions specified in the protocol
* Negative drug screen

Exclusion Criteria:

* Participation in another clinical trial in the last 3 months
* Significant allergies, allergic diathesis or known hypersensitivity for ketamine or its ingredients (ie, Benzethonium chloride)
* History of or current significant respiratory disease, cardiovascular disease, endocrinological, gastrointestinal, neurological, glaucoma and known liver and kidney failure
* Contraindications for an MRI being performed (claustrophobia, metal parts, pacemaker)
* oxygen saturation pO2 < 90 mmHg
* Clinically significant abnormalities in ECG or laboratory values
* Recent history (within previous 6 months) of alcohol or drug abuse
* History of or current psychiatric diagnoses (DSM-IV, II) or neurological disorders
* Relatives in first or second degree with a schizophrenic disorder
* Serology positive for hepatitis B surface antigen, hepatitis C antibodies or HIV antibodies
* Signs of hyperthyroidism based on the determination of T3, T4 and TSH

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-10; Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Cerebral activation of ketamine as determined by functional MRI | 25 and 40 minutes after end of bolus injection of ketamine/placebo
Cerebral activation of ketamine as determined by electroencephalogram (EEG) during an oddball-task | 25 and 40 minutes after end of bolus injection of ketamine/placebo

SECONDARY OUTCOMES:
Effect of Ketamine on consciousness as measured by the "Altered States of Consciousness Rating Scale" | 60 min after end of bolus injection of ketamine.
Cerebral activation induced by ketamine as measured by simultaneous fMRI / EEG under resting conditions | 0 and 25 min after end of bolus injection of ketamine.
Symptom score of ketamine as measured with the Positive And Negative Symptom Scale | 60 min after end of bolus injection of ketamine (= at the end of ketamine infusion).

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.